CLINICAL TRIAL: NCT06114147
Title: Cardiac Flow Measurements in Pregnant Women by Non Invasive Techniques: Comparison Between USCOM, ICON and Trans Thoracic Echography
Brief Title: Cardiac Flow Measurements in Pregnant Women by Non Invasive Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Bénédicte LE TINIER, doctor in medecine,assistant to the head of department in charge of the antenatal consultation unit, principal investigator, University of Geneva, Switzerland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-D0100
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Pregnancy Related; Cardiac Output

STUDY DESIGN:
Intervention Model Description: prospective cross sectional study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- pregnant women (Experimental): pregnant women with eligibility criteria with gestational age from 12 to 16+6/7 WA and then from 32 to 36+6/7 WA.
  Interventions: Device: trans thoracic echocardiography measure; Device: ICON measure; Device: USCOM

INTERVENTIONS:
Device: trans thoracic echocardiography measure — The trans thoracic echography would be carried out with cardiac classic sections to ensure the structural cardiac and valvular normality and then sections repeated 3 times over 10 minutes will be carried out to calculate the cardiac output.
Device: ICON measure — The ICON will be placed at the beginning of the consultation and the measurements will be taken at the same time as the trans thoracic ultrasound in the left lateral decubitus position.
Device: USCOM — Afterwards, measurements will be made with USCOM in left lateral position and 3 of the best spectra archived according to the Fremantle score.

SUMMARY:
the goal of this clinical trial is to compare the measurement of cardiac output, systolic ejection volume and vascular filling in pregnant women with the new non-invasive measurement techniques of the Index of contractility monitor (ICON) and the Ultra Sonic Cardiac Output Monitor (USCOM) in pregnant women compared to trans-thoracic ultrasound as the gold standard of non-invasive techniques The Secondary objective is to evaluate patient comfort between the 3 techniques, examination time and examiner satisfaction.

The main question it aim to answer is the absence or a low difference in cardiac output measurement ( less than 30 %) between the non invasive measurement methods ( USCOM/ICON) and the trans thoracic cardiac echography in pregnant women in the first and third trimester.

DETAILED DESCRIPTION:
It is a Prospective cross sectional study

The study design does not allow for randomisation or double-blinding.

Patients will be enrolled in the first trimester of pregnancy and offered the study at the 10 gestational week (GW) consultation. After signing and giving informed consent, the research nurse or midwife will schedule the specific consultation from between 12 to and 16+6 Weeks of Amenorrhea (WA) (cardiac output rise from 5 weeks of gestation to 16 weeks of gestation and then stay at the same level) and in the 3rd trimester from between 32 to and 36+6 WA. Patients will therefore be included from the beginning of their pregnancy until their delivery, i.e. approximately 7 months All pregnant patients will each have a measurement in left lateral decubitus by the 3 devices from 12 to 16+6 WA and another set of measurement between 32 and 36+6 WA.

During the specific consultations organized (eg on Tuesday mornings), a designed medical professional will carry out measurement with the 3 different devices in a room accordingly with an examination table allowing the left lateral decubitus. At each consultation parameters such as weight, height of the patient, cardiac frequency, blood pressure will be recorded.

Each consultation is expected to last 30 minutes: The ICON will be placed at the beginning of the consultation and the measurements will be taken at the same time as the trans thoracic ultrasound in the left lateral decubitus position. The trans thoracic echography would be carried out with cardiac classic sections to ensure the structural cardiac and valvular normality and then sections repeated 3 times over 10 minutes will be carried out to calculate the cardiac output. Afterwards, measurements will be made with USCOM in left lateral position and 3 of the best spectra archived according to the Fremantle score.

The person performing the measurements will be an ultrasound laboratory technician trained in trans thoracic echocardiography according to Cardiology societies recommendations that consider that three months of full-time experience and 150 echocardiograms are required to be fully competent in echocardiography.

For measurements with USCOM and ICON, the technician will have an adequate training beforehand to formalize with the 2 devices and then perform the measurements during the dedicated consultations. The images for each measurement selected with each device will be stored on a USB key for USCOM and ICON and then transferred to KHEOPS by the research midwife respecting anonymization using the study number attributed for each patient. For the transthoracic ultrasound, the interest of the patient is paramount, these images will be transferred from the ultrasound machine to the secure server of the Universitary Hospital of Geneva (HUG) with the patient's identity and can be annexed to the integrated patient medical file so that these images can be used as a comparison in case of later consultation for cardiac symptoms. The images will be analyzed by the cardiologist investigator in the study who will have access to a secure database with patient identity and patient's study number so as to recover the cardiac images. He will calculate the cardiac output according to the following formula: the Cardiac output can be calculated after measuring the systolic ejection volume at the aortic annulus. At this level, the diameter of the annulus is measured during systole using two-dimensional ultrasound. Subsequently, the time-velocity integral of aortic ejection (VTIao) can be obtained using pulsed Doppler at the annulus. The systolic ejection volume is equal to the product of VTIao the diameter of the annulus squared multiplied by divided by 4 (VES = VTIao x ( D2/4) and the cardiac output will be equal to this value multiplied by the heart rate during measurement.

At the end of each examination, the laboratory technician will rate the objective values for each of the 2 devices: duration of the examination to obtain an interpretable measurement measured by a stopwatch that is started and then stopped when the measurement is performed in a satisfactory manner for the operator. Subjective values such as the feeling of comfort will be asked for each examination to the patient before moving on to the next examination according to a simple verbal scale : comfortable/ uncomfortable/ unbearable to be ticked on redcap. At the end of the consultation, the operator will assess the ease of measurement with the 3 devices using a simple verbal scale :easy/ moderately easy/ moderately difficult/ difficult to be ticked on redcap.

The measurement values for USCOM and ICON will be entered into redcap at the end of each consultation by the research midwife from the data on the USB ( Universal serial bus) stick transferred into KHEOPS software. The patient's medical data will be completed in redcap by the research midwife from the integrated patient record. The cardiac output measurement will be performed by the study cardiologist from the images transferred to the patient's integrated file (DPI) under the patient's identity and reopened thanks to the secure database associating the patient's identity and the unique study number accessible only to the investigators. The principal investigator and the statistician will interpret the anonymized raw data and will not be involved in the measurements. Due to the comparison of 3 devices easily recognizable by their shape, the study will be an open study. The stored images will be reviewed to ensure the quality of the Doppler spectrum for USCOM according to the Fremantle score and the measurement of cardiac output with transthoracic ultrasound at the level of the aortic valve. The Fremantle score is used to check the quality of the USCOM spectrum. The expected score for a good USCOM spectrum is 6. A score < 4 defines an insufficient spectrum quality. The echocardiography measurements will be used as a comparison as it is considered the gold standard for non-invasive cardiac output measurement.

The investigators need to include 100 patients by recruiting them in the first trimester of pregnancy and they will remain included until delivery. Some pregnancies may develop complications preventing from having the second measurement from 32 to 36 WA. The investigators need to obtain 100 measurements from 12 to 16 WA and 100 from 32 to 36 WA. The investigators will therefore have to re-include as many patients from 32 to 36 WA as those who gave birth before this 3rd trimester measurement. So this number of 100 patients can be more to obtain 100 measures at first trimester and 100 measures at third trimester. As investigators are comparing devices and the ease of use of these devices, without correlating the data to a clinical outcome, not having continuity between patients in the first and third trimester does not constitute a bias.

The duration of the project will be 18 months to obtain 100 measurements with the 3 devices from 12 to 16 WA and 100 measurements in the 3rd trimester of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Any pregnant person over 16 years old followed at the prenatal consultation of the maternity ward of the Geneva University Hospitals.

Exclusion Criteria:

* Drug or alcohol abuse,
* Miscarriage or intra uterine demise before the first exam.
* Inability to follow the procedures of the investigation, e.g. due to psychological disorders, dementia, etc. of the subject,
* Inability to give an informed consent.
* preexisting or congenital cardiopathy
* Structural abnormalities of hearth or valves diagnosed in the first Trans Thoracic Echocardiography screening

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
difference in cardiac output | 18 month
  Absence/low difference in cardiac output measurement (less than 30% difference) between the new non-invasive measurement methods (USCOM, ICON) and the trans thoracic echocardiography in pregnant women in the first and third trimester of pregnancy compared to the reference method which is trans thoracic echocardiography.

SECONDARY OUTCOMES:
stroke volume | 18 month
  To compare the stroke volume of USCOM and ICON to trans thoracic echocardiography between USCOM and ICON.
systemic vascular resistance | 18 month
  To compare the systemic vascular resistance between USCOM and ICON.
patient satisfaction | 18 month
  measure with a verbal scale of 3 choices : comfortable, uncomfortable, insupportable for each measurement
user satisfaction | 18 month
  measure with a verbal scale of 4 choices: easy, moderately easy, moderately difficult, difficult for each measurement
examination time | 18 month
  Examination time in minutes for each measurement

CONTACTS AND LOCATIONS:
Overall Officials: Bénédicte LE TINIER, MD, Principal Investigator — Hopitaux universitaires de Geneve
Locations (1):
- Hopitaux Universitaires de Geneve, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No